CLINICAL TRIAL: NCT07296809
Title: A Phase II, Multicenter, Open-Label Study to Evaluate the Safety and Efficacy of SKB500 Combinations in Patients With Small Cell Lung Cancer
Brief Title: SKB500 Combinations in Patients With Small Cell Lung Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sichuan Kelun-Biotech Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Sichuan Kelun Pharmaceutical Research Institute Co., Ltd. (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SKB500-II-02
Record Dates: First submitted 2025-11-25; First posted 2025-12-22 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Small Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Injections; 18-O-demethylcervinomycin A2; Carboplatin; Etoposide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 1. SKB500+KL-A167 (Experimental): Participants will receive KL-A167 followed by SKB500
  Interventions: Drug: SKB500 Powder for Injection; Drug: KL-A167 Injection
- 2. SKB500 +KL-A167+Carboplatin (Experimental): Participants will receive KL-A167 followed by SKB500 with Carboplatin
  Interventions: Drug: SKB500 Powder for Injection; Drug: KL-A167 Injection; Drug: Carboplatin Injection
- 3. SKB500+KL-A167+Carboplatin+Etoposide (Experimental): Participants will receive KL-A167 followed by SKB500, Carboplatin with Etoposide
  Interventions: Drug: SKB500 Powder for Injection; Drug: KL-A167 Injection; Drug: Carboplatin Injection; Drug: Etoposide Injection

INTERVENTIONS:
Drug: SKB500 Powder for Injection — SKB500 will be administered as an intravenous (IV) infusion, every 3 weeks on Day 1 of each 21-day cycle and the dose will be determined based on the efficacy and safety data from the SKB500-I-01 study.
Drug: KL-A167 Injection — KL-A167 will be administered as an intravenous (IV) infusion every 3 weeks on Day 1 of each 21-day cycle (1200mg)
Drug: Carboplatin Injection — Carboplatin will be administered as an intravenous (IV) infusion every 3 weeks on Day 1 of each 21-day cycle（AUC 5, Cycles 1-4)
  Arms: 2. SKB500 +KL-A167+Carboplatin; 3. SKB500+KL-A167+Carboplatin+Etoposide
Drug: Etoposide Injection — Etoposide will be administered as an intravenous (IV) infusion every 3 weeks on Day 1, 2, and 3 of each 21-day cycle (100 mg/m^2, Cycles 1-4).
  Arms: 3. SKB500+KL-A167+Carboplatin+Etoposide

SUMMARY:
The purpose of this study is to assess the safety, tolerability and preliminary antitumor activity of SKB500 combinations in patients with small cell lung cancer. The study is divided into two parts. Part 1 will be the safety run-in phase, and Part 2 will be the cohort expansion phase.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants between 18 and 75 years old.
2. Histologically or cytologically confirmed Extensive-stage small cell lung cancer (ES-SCLC):

   * Cohort 1: participant has received or not received prior systemic treatment, with no more than 1 prior systemic therapy in the extensive stage.
   * Cohort 2~3: participant has received no prior systemic treatment.
3. Agree to provide fresh or archival tumor tissue for biomarker analysis.
4. Has at least one measurable lesion according to Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1.
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
6. Life expectancy >= 12 weeks.
7. Has adequate organ and bone marrow functions.
8. Has recovered to grade ≤ 1 of prior anti-cancer treatment toxicities.
9. Effective contraceptive methods should be used during the study and for 6 months after the end of treatment.
10. Voluntarily join this study, sign the informed consent form, and can comply with the protocol-specified visits and procedures.

Exclusion Criteria:

1. The pathology suggests the presence of both non-small cell carcinoma and small cell carcinoma components.
2. Has previously received medications with the same target or the same toxins.
3. Presence of spinal cord compression or clinically active central nervous system metastases.
4. Presence of clinical symptoms caused by tumor invasion or compression of important organs and blood vessels.
5. Severe infection within 4 weeks or active infection requiring systemic anti-infective treatment within 2 weeks prior to the first dose.
6. With peripheral neuropathy of grade ≥ 2.
7. History of any serious, life threatening, or permanently discontinuing adverse events mediated by immunotherapy, including infusion reactions.
8. Presence of uncontrolled concurrent diseases, including but not limited to decompensated liver cirrhosis, nephrotic syndrome, uncontrolled metabolic disorders, Severe active peptic ulcer, gastrointestinal bleeding, gastrointestinal perforation, intestinal obstruction, etc.
9. Serious or uncontrolled heart disease or clinical symptoms requiring treatment.
10. History of interstitial lung disease (ILD) /noninfectious pneumonitis that require steroid treatment, or currently has ILD/noninfectious pneumonitis.
11. Clinical severe lung damage caused by concurrent lung disease.
12. Uncontrolled hypertension, diabetes, or repeated drainage of pleural effusion/pericardial effusion/ abdominal effusion.
13. Pregnant or lactating women.
14. Rapid disease deterioration in the screening process.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-12-20 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events (AEs) | up to 24 months
  Incidence and severity of adverse events (AEs) graded by Common Terminology Criteria for Adverse Events (CTCAE) v5.0
Progression-free survival (PFS) | up to 24 months
  Progression-free survival (PFS) was defined as the time from baseline to the earliest date of the first objective documentation of progressive disease (PD) or death due to any cause.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | up to 24 months
  Objective Response Rate (ORR) is the percentage of participants who achieved a best overall response of Complete Response (CR) or Partial Response (PR), assessed by Investigator based on RECIST version 1.1.
Duration of response (DOR) | up to 24 months
  Duration of Response (DOR) was defined as the time from the date of the first documentation of objective response (complete response [CR] or partial response [PR]) to the date of the first objective documentation of progressive disease (PD) or death due to any cause. DoR was measured for responding subjects (PR or CR) only.
Disease control rate (DCR) | up to 24 months
  Disease control rate (DCR) was defined as the sum of complete response (CR) rate, partial response (PR) rate, and stable disease (SD) rate. As per RECIST v1.1, CR was defined as a disappearance of all lesions, PR was defined as at least a 30% decrease in the sum of diameters of target lesions, and stable disease (SD) was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease.
Overall Survival (OS) | up to 24 months
  The time from first dose to death from any cause.
Pharmacokinetic Parameter Maximum Plasma Concentration (Cmax) of SKB500-ADC, SKB500-TAB and free payload | Cycle 1-4, 6, 8,12,16, every 8 cycles starting from Cycle 16 Day 1: pre-dose, post-dose (each cycle is 21 days), up to 24 months
Pharmacokinetic Parameter Minimum Plasma Concentration (Cmin) of SKB500-ADC, SKB500-TAB and free payload | Cycle 1-4, 6, 8,12,16, every 8 cycles starting from Cycle 16 Day 1: pre-dose, post-dose (each cycle is 21 days), up to 24 months, up to 24 months
Anti-drug Antibodies (ADA) for SKB500 | Cycle 1-4, 6, 8, 12, 16, every 8 cycles starting from Cycle 16 Day 1: pre-dose, (each cycle is 21 days), up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Yilong Wu, Principal Investigator — Guangdong Provincial People's Hospital
Locations (1):
- Guangdong Provincial People's Hospital, Guangzhou, Guangdong, China